CLINICAL TRIAL: NCT07387510
Title: A Phase Ⅱ, Single-arm, Open-label Trial of DGPR1008 for Intraoperative Fluorescence Imaging of Prostate-specific Membrane Antigen-positive Prostate Cancer
Brief Title: PSMA-Targeted Intraoperative Fluorescent Imaging Agents (DGPR1008): Validation Across Different Time Windows
Acronym: DGPR1008-04
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haitao Niu, MD (Other)
Responsible Party: Sponsor-Investigator, Haitao Niu, MD, Clinical Professor, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2026-009-01
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): DGPR1008 (0.04 mg/kg according to each subject's body weight) was given as a single slow infusion 12 hours (±4 hours) preoperatively, after which radical prostatectomy was performed. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Interventions: Drug: 12 h before RP
- group 2 (Experimental): DGPR1008 (0.04 mg/kg according to each subject's body weight) was given as a single slow infusion 24 hours (±4 hours) preoperatively, after which radical prostatectomy was performed. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Interventions: Drug: 24 h before RP
- group 3 (Experimental): DGPR1008 (0.04 mg/kg according to each subject's body weight) was given as a single slow infusion 36 hours (±4 hours) preoperatively, after which radical prostatectomy was performed. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Interventions: Drug: 36 h before RP

INTERVENTIONS:
Drug: 12 h before RP — DGPR1008 (0.04 mg/kg according to each subject's body weight) was given as a single slow infusion 12 hours (±4 hours) preoperatively, after which radical prostatectomy was performed. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Arms: group 1
Drug: 24 h before RP — DGPR1008 (0.04 mg/kg according to each subject's body weight) was given as a single slow infusion 24 hours (±4 hours) preoperatively, after which radical prostatectomy was performed. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Arms: group 2
Drug: 36 h before RP — DGPR1008 (0.04 mg/kg according to each subject's body weight) was given as a single slow infusion 36 hours (±4 hours) preoperatively, after which radical prostatectomy was performed. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Arms: group 3

SUMMARY:
a Phase II, single-arm, open-label, multi-center study to evaluate safety, tolerability, pharmacokinetics, and the effectiveness of near-infrared fluorescence imaging during surgery.

DETAILED DESCRIPTION:
We plan to enroll 27 prostate cancer patients and divide them into 3 different time-window groups. Intravenous administration will be conducted 12/24/36 hours before surgery. Blood samples will be collected for relevant tests, and fluorescence imaging will be performed during the operation. After surgery, the intraoperative imaging results will be compared with pathological findings to draw relevant conclusions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with prostate cancer through preoperative transrectal prostate biopsy and pathological examination, who are scheduled to undergo radical prostatectomy with or without pelvic lymph node dissection;
2. Subjects must provide informed consent prior to trial initiation, fully understand the trial content, procedures, and potential adverse reactions, be capable of effective communication with the investigator, and be able to complete the trial as per protocol requirements. They must voluntarily sign a written informed consent form;
3. Adult male subjects aged 18 years or older (including the boundary value);
4. Gleason score ≥7, or imaging studies (transrectal ultrasound [TRUS] and/or prostate magnetic resonance imaging [MRI] or CT or PSMA PET/CT) demonstrating disease staging ≥T2, or imaging evidence of regional lymph node enlargement suggestive of lymph node metastasis;
5. No hepatic or renal impairment: Hepatic: Total bilirubin ≤ 2 times the upper limit of normal (ULN) (excluding Gilbert syndrome), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3×ULN; Renal: Creatinine clearance ≥ 50 mL/min/1.73 m² (simplified MDRD formula);
6. The investigator determines the subject has no clear contraindications for surgery and is suitable for radical prostatectomy;
7. The subject and their partner or spouse must agree to have no plans for pregnancy or sperm donation from the screening period until 3 months after trial completion, and voluntarily use effective contraception.

Exclusion Criteria:

Subjects will be excluded if they meet any one of the following criteria:

1. Subjects with a history of allergies (e.g., known allergies to two or more medications), those prone to allergic reactions such as rashes or hives, or those with known allergies to the investigational drug (including its formulation components);
2. Subjects with significantly abnormal screening test results deemed clinically significant by the investigator and likely to affect study participation; or those with concomitant conditions posing serious safety risks or impeding study completion (except where the investigator determines the condition is stable and allows enrollment);
3. Subjects who participated in another clinical trial involving investigational drugs or devices within the month preceding study drug administration;
4. Subjects who have undergone neoadjuvant therapy, radiation therapy, focal ablation therapy, hormone therapy, or androgen deprivation therapy within the past 6 months;
5. Subjects deemed by the investigator to have other conditions rendering them unsuitable for participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-07-27 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of DGPR-1008 (administered 12 hours prior) in conjunction with a near-infrared fluorescence imaging device for intraoperative detection in patients. | From the screening period to the Day 7 of the trial
  Detection of prostate cancer tissue by DGPR1008 using near-infrared fluorescence (NIR) imaging at 12 hours after intravenous administration to subjects. Evaluate the sensitivity (or true positive rate, TP/[TP+FN]), specificity (or true negative rate, TN/[TN+FP]), false positive rate (FP/[FP+TN]), and false negative rate (FN/[FN+TP]) of DGPR-1008 for detecting prostate cancer tissue in near-infrared fluorescence imaging (NIR) during radical prostatectomy. The proportion of additionally resected tissues that are diagnosed as tumors by pathological evaluation.
Evaluate the efficacy of DGPR-1008 (administered 24 hours prior) in conjunction with a near-infrared fluorescence imaging device for intraoperative detection in patients. | From the screening period to the Day 7 of the trial
  Detection of prostate cancer tissue by DGPR1008 using near-infrared fluorescence (NIR) imaging at 24 hours after intravenous administration to subjects. Evaluate the sensitivity (or true positive rate, TP/[TP+FN]), specificity (or true negative rate, TN/[TN+FP]), false positive rate (FP/[FP+TN]), and false negative rate (FN/[FN+TP]) of DGPR-1008 for detecting prostate cancer tissue in near-infrared fluorescence imaging (NIR) during radical prostatectomy. The proportion of additionally resected tissues that are diagnosed as tumors by pathological evaluation.
Evaluate the efficacy of DGPR-1008 (administered 36 hours prior) in conjunction with a near-infrared fluorescence imaging device for intraoperative detection in patients. | From the screening period to the Day 7 of the trial
  Detection of prostate cancer tissue by DGPR1008 using near-infrared fluorescence (NIR) imaging at 36 hours after intravenous administration to subjects. Evaluate the sensitivity (or true positive rate, TP/[TP+FN]), specificity (or true negative rate, TN/[TN+FP]), false positive rate (FP/[FP+TN]), and false negative rate (FN/[FN+TP]) of DGPR-1008 for detecting prostate cancer tissue in near-infrared fluorescence imaging (NIR) during radical prostatectomy. The proportion of additionally resected tissues that are diagnosed as tumors by pathological evaluation.

SECONDARY OUTCOMES:
Evaluate DGPR1008 combined with near-infrared fluorescence imaging devices for detecting positive margins in histopathological examination following radical prostatectomy | From the screening period to the Day 7 of the trial
  To evaluate the proportion of subjects with a positive surgical margin (PSM) score of ≥1, as assessed by histopathology, at different time points after radical prostatectomy.
Evaluate DGPR1008 combined with near-infrared fluorescence imaging devices for detecting positive lymph nodes in histopathological examination following radical prostatectomy | From the screening period to the Day 7 of the trial
  To evaluate the proportion of subjects with positive lymph nodes, as assessed by histopathology, at different time points after radical prostatectomy.
Evaluate the safety of single-dose administration of DGPR1008 in patients | From the screening period to the Day 7 of the trial
  Adverse event collection, including (such as the location, nature, and frequency of pain), physical signs (such as the scope of rash, blood pressure values), laboratory abnormal values and units (such as ALT 200 U/L), etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF